CLINICAL TRIAL: NCT02557594
Title: A Randomized, Open-label, Two-way Crossover Study to Assess the Safety and Pharmacokinetics of DA-2802 319mg and Viread 300mg After a Single Oral Dose in Healthy Male Volunteers
Brief Title: Clinical Trial to Assess the Safety and Pharmacokinetics of DA-2802 319mg and Viread 300mg in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA2802_BE_I
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viread → DA-2802 (Experimental): * Viread 300mg(Tenofovir disoproxil fumarate)
  * DA-2802 319mg(Tenofovir disoproxil orotate)
  Interventions: Drug: Viread 300mg; Drug: DA-2802 319mg
- DA-2802 → Viread (Experimental): * Viread 300mg(Tenofovir disoproxil fumarate)
  * DA-2802 319mg(Tenofovir disoproxil orotate)
  Interventions: Drug: Viread 300mg; Drug: DA-2802 319mg

INTERVENTIONS:
Drug: Viread 300mg — single dose administration after 10hr fasting
  Other Names: Tenofovir disoproxil fumarate
Drug: DA-2802 319mg — single dose administration after 10hr fasting
  Other Names: Tenofovir disoproxil orotate

SUMMARY:
This Phase I clinical study is to evaluate the safety and pharmacokinetics of DA-2802 319mg and Viread 300mg after a single oral dose in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 50, healthy male subjects(at screening)
* Body weight over 55kg, BMI between 18.0 - 27.0
* Volunteer who totally understands the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Volunteer who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, neurology, immunology, pulmonary, endocrine, hematooncology, urinary, skeletomuscular, cardiovascular, mental disorder)
* Volunteer who had GI tract disease(Crohn's disease, ulcer, acute or chronic pancreatitis) or surgery(appendectomy, hernioplasty are excluded)
* Genetic disorders such as glucose-galactose malabsorption, Lapp lactose deficiency, galactose intolerance which is contraindication to Viread
* Volunteer who had hypersensitivity reaction to medicines including Tenofovir, Aspirin, or antibiotics
* exceed 1.5 times the normal range of AST, ALT at screening test before randomization
* history of drug abuse, or a positive urine drug screen
* having ETC drug or herbal medicines within 2 weeks before first administration or OTC drug or vitamin preparations within a week before first administration
* Participation in any other clinical trial involving investigational drugs within 3 months
* Volunteer who had whole blood donation in 2 months, or component blood donation or transfusion in 1 months
* Regular alcohol consumption(over 21 units/week, 1unit=10g of pure alcohol) or volunteers who cannot abstain from drinking during the study
* Volunteers smoking over 10 cigarettes per day or who cannot abstain from smoking during the study(from 24hr before admission to discharge)
* Volunteers who had grapefruit containing foods from 24hr before admission to discharge or who cannot abstain from grapefruit containing foods
* Volunteers who are not using adequate contraception methods or have a pregnancy plan
* volunteers who cannot abstain from caffeine containing foods(coffee, tea, soft drinks etc) during the study
* any condition that, in the view of the investigator, would interfere with study participation

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2016-03-08 (Actual)

PRIMARY OUTCOMES:
Area Under Curve(AUC)last of Tenofovir | 0h(before admisitration), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72h post-dose
Maximum of concentration(Cmax) of Tenofovir | 0h(before admisitration), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72h post-dose

SECONDARY OUTCOMES:
Time of maximum concentration(Tmax) of Tenofovir | 0h(before admisitration), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72h post-dose
Terminal half-life(t1/2) of Tenofovir | 0h(before admisitration), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72h post-dose
Apparent Clearance(CL/F) of Tenofovir | 0h(before admisitration), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72h post-dose
Area Under Curve(AUC)inf of Tenofovir | 0h(before admisitration), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, Ph.D, M.B.A, Principal Investigator — Seoul National University Hospital
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea